CLINICAL TRIAL: NCT07318493
Title: Does Antiseptic Coated Suture Reduce Pancreatic Fistula Rate After Pancreatoduodenectomy: A Randomized Controlled Trial
Brief Title: Antiseptic-Coated Sutures and Pancreatic Fistula Risk After Pancreatoduodenectomy
Acronym: Triclosan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, Toms Augustin, Medical Director (Main Campus) - Safety, Quality and Patient Experience, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-575
Record Dates: First submitted 2025-11-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pancreatoduodenectomy; Whipple Procedure
Keywords: pancreatoduodenectomy; whipple procedure; sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard (non-antiseptic coated) suture will be used. (Other): You will undergo your primary surgery per standard practice at the discretion of your surgeon. Standard Sutures will be used during your operation.
  Interventions: Device: Standard (non-antiseptic coated) suture will be used.
- Triclosan/antiseptic -coated suture (Other): You will undergo your primary surgery per standard practice at the discretion of your surgeon. Triclosan/antiseptic -coated suture will be used. Ethicon PDSTM Plus Antibacterial Suture will be used at the layer of the pancreatojejunostomy and for the duration of the case.
  Interventions: Device: Triclosan/antiseptic -coated suture

INTERVENTIONS:
Device: Standard (non-antiseptic coated) suture will be used. — This is an operation to treat tumors and other conditions in the pancreas, small intestine, and bile ducts. It involves removing the head of the pancreas, the first part of the small intestine, the gallbladder, and the bile duct. Part of the procedure involves sutures. A suture(s) is a stitch or row of stitches holding together the edges of a wound or surgical incision
  Arms: Standard (non-antiseptic coated) suture will be used.
Device: Triclosan/antiseptic -coated suture — Triclosan/antiseptic -coated suture will be used. Ethicon PDSTM Plus Antibacterial Suture will be used at the layer of the pancreatojejunostomy and for the duration of the case.
  Arms: Triclosan/antiseptic -coated suture

SUMMARY:
The purpose of this study is to determine if the use of antiseptic-coated sutures is better than the use of the standard sutures in preventing postoperative fistulas within 90 days after pancreatoduodenectomy.

DETAILED DESCRIPTION:
This study is a randomized-controlled trial comparing the rate of post-operative pancreatic fistula (POPF) in patients undergoing pancreatoduodenectomy. This is a superiority study designed to determine whether the use of antiseptic-coated sutures (intervention arm) is superior to standard sutures (control arm) in regard to clinically significant POPF within 90 days following pancreatoduodenectomy. Patients will be randomized to receive either a pancreatoduodenectomy surgery utilizing antiseptic coated sutures or with non-coated standard sutures. The study hypothesize that the use of antiseptic-coated sutures will be associated with a reduction in the rate of POPF. Both sutures are currently available at our center and utilized in the procedure of interest.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be undergoing a scheduled pancreatoduodenectomy.
* Age ≥18 years.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients < 18 years old
* Patients who are pregnant
* Patients with history of previous pancreatic surgery
* Patients who are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of the rate of postoperative pancreatic fistula | up to 90 days post-operative
  comparison of the rate of postoperative pancreatic fistula- Biochemical leak
Comparison of the rate of postoperative pancreatic fistula | up to 90 days post-operative
  Comparison of the rate of postoperative pancreatic fistula-Grade B
Comparison of the rate of postoperative pancreatic fistula | up to 90-day post operative
  Comparison of the rate of postoperative pancreatic fistula-Grade C

SECONDARY OUTCOMES:
Improvement in Rate of clinically significant POPF | up to 90-days post-operative
  Improvement in Rate of clinically significant POPF (Grade B and C defined by ISGLS definition)
Improvement in SSI rates between groups using CDC classification | up to 90-days post-operative
  Improvement in SSI rates between groups using CDC classification (superficial, deep, organ space)
Hospital Length of Stay | up to 90-day post operative
  Duration of hospital admission, measured in days, during index presentation for pancreatoduodenectomy. This will subsequently be compared among our two cohorts (standard suture vs antiseptic suture)
Length of ICU stay | up to 90-day post operative
  Duration of Intensive care unit admission, measured in days, during index presentation for pancreatoduodenectomy, or during convalescence from surgery. This will subsequently be compared among our two cohorts (standard suture vs antiseptic suture)
Surgical Site Infection | up to 90-day post operative
  An infection that occurs in the part of the body where the surgery took place and includes superficial, deep, and organ space infections
Surgical site occurrence | Up to 90 days post-operative
  Non-healing incisional wound, fascial disruption, skin or soft tissue ischemia, skin or soft tissue necrosis, wound serous or purulent drainage, stitch abscess, seroma, hematoma, wound dehiscence, and enterocutaneous fistula
Surgical Site Occurrence requiring Procedural Intervention | up to 90 days post-operative
  Interventions to address wound healing issues or complications including wound opening or debridement, suture excision, percutaneous drainage. This includes to address superficial, deep, and organ space healing concerns
Post operative pancreatic fistula interventions | Up to 90 days post-operative
  Postoperative interventions related to clinically relevant postoperative pancreatic leak (defined by 2016 International Study Group of Pancreatic Fistula) including percutaneous, endoscopic and surgical interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Toms Augustin, MD, Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (3):
  - Cleveland Clinic Akron, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Cleveland Clinic Fairview Hospital, Fairview, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shubert CR, Wagie AE, Farnell MB, Nagorney DM, Que FG, Reid Lombardo KM, Truty MJ, Smoot RL, Kendrick ML. Clinical Risk Score to Predict Pancreatic Fistula after Pancreatoduodenectomy: Independent External Validation for Open and Laparoscopic Approaches. J Am Coll Surg. 2015 Sep;221(3):689-98. doi: 10.1016/j.jamcollsurg.2015.05.011. Epub 2015 May 21. PMID 26296680
- [Background] Shubert CR, Kendrick ML, Habermann EB, Glasgow AE, Borah BJ, Moriarty JP, Cleary SP, Smoot RL, Farnell MB, Nagorney DM, Truty MJ, Que FG. Implementation of prospective, surgeon-driven, risk-based pathway for pancreatoduodenectomy results in improved clinical outcomes and first year cost savings of $1 million. Surgery. 2018 Mar;163(3):495-502. doi: 10.1016/j.surg.2017.10.022. Epub 2017 Dec 21. PMID 29275974
- [Background] Ocuin LM, Loftus A, Elshami M, Hue JJ, Musonza T, Ammori JB, Winter JM, Hardacre JM. Extended antibiotic therapy is associated with a lower rate of clinically relevant postoperative pancreatic fistula after pancreatoduodenectomy in intermediate- and high-risk patients: A single-institution analysis. Surgery. 2024 Feb;175(2):477-483. doi: 10.1016/j.surg.2023.09.049. Epub 2023 Nov 7. PMID 37940433
- [Background] Riall TS, Nealon WH, Goodwin JS, Townsend CM Jr, Freeman JL. Outcomes following pancreatic resection: variability among high-volume providers. Surgery. 2008 Aug;144(2):133-40. doi: 10.1016/j.surg.2008.03.041. PMID 18656618
- [Background] Krautz C, Nimptsch U, Weber GF, Mansky T, Grutzmann R. Effect of Hospital Volume on In-hospital Morbidity and Mortality Following Pancreatic Surgery in Germany. Ann Surg. 2018 Mar;267(3):411-417. doi: 10.1097/SLA.0000000000002248. PMID 28379871
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Yang YM, Tian XD, Zhuang Y, Wang WM, Wan YL, Huang YT. Risk factors of pancreatic leakage after pancreaticoduodenectomy. World J Gastroenterol. 2005 Apr 28;11(16):2456-61. doi: 10.3748/wjg.v11.i16.2456. PMID 15832417
- [Background] Sato N, Yamaguchi K, Chijiiwa K, Tanaka M. Risk analysis of pancreatic fistula after pancreatic head resection. Arch Surg. 1998 Oct;133(10):1094-8. doi: 10.1001/archsurg.133.10.1094. PMID 9790207